CLINICAL TRIAL: NCT03492333
Title: The Role of Antigliadin Antibodies in Predicting the Beneficial Effect of Gluten Free Diet in Unselected IBS Patients
Brief Title: Gluten Free Diet in IBS Patients Stratified According to Their Antigliadin Status
Acronym: GFD_IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AGA_GFD_in_IBS
Record Dates: First submitted 2018-04-03; First posted 2018-04-10 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2017-07

CONDITIONS: IBS - Irritable Bowel Syndrome
Keywords: antigliadin, gluten free diet, transit
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Diet, Gluten-Free

STUDY DESIGN:
Intervention Model Description: Intervention GFD in IBS and HV(controls)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gluten free diet (Experimental): Single arm
  Interventions: Other: Gluten free diet

INTERVENTIONS:
Other: Gluten free diet — Gluten-free diet- Instructions provided by a dietitian

SUMMARY:
Gluten-free diet has been shown to improve gut symptoms in patients with celiac disease and also in adult patients with diagnosis of Irritable Bowel Syndrome (Rome III criteria).

Antibodies to native gliadin (AGA) have been suggested as a potential diagnostic marker of response to GFD. However, this has not been tested in a prospective study in IBS patients. Identification of predictors of a symptomatic response to GFD within the IBS population would improve the clinical management of these patients.

The purpose of this study is to evaluate the effect of gluten-free diet on gastrointestinal symptoms and gut motility in patients with Irritable Bowel Syndrome stratified according to their antigliadin antibodies status.

Additional purposes include investigating effects gluten free diet may have on other parameters:

* Improvement of mood
* Quality of life and general well-being
* Changes in gut microbiota

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* IBS diagnosis (Rome III)
* Willingness to participate

Exclusion Criteria:

* history of any organic disease including celiac disease
* Immune deficiency
* Major abdominal surgery
* Use of immunosuppressants, glucocorticosteroids or opioids
* Use of antibiotics in the last 3 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2012-04-30 (Actual); Primary Completion 2016-05-30 (Actual); Study Completion 2016-05-30 (Actual)

PRIMARY OUTCOMES:
Improvement on gastrointestinal symptoms | 4 weeks
  Decrease >2 points IBS Birmingham score

SECONDARY OUTCOMES:
Normalization of gastrointestinal transit | 4 weeks
  (SHAPE 25-50 radiopaque markers)
Improvement anxiety and/or depression | 4 weeks
  Decrease >2 points Hospital anxiety and depression (HAD) score
Improvement somatization | 4 weeks
  Decrease somatization scores (PHQ15)
Improvement quality of life and well-being | 4 weeks
  Decrease in the psychological general well-being (PGWB) score
Changes in gut microbiota | 4 weeks
  changes in microbial composition

CONTACTS AND LOCATIONS:
Overall Officials: Premysl Bercik, MD, Principal Investigator — McMaster University
Locations (1):
- Farncombe Institute, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No plan to share data.

REFERENCES:
- [Derived] Pinto-Sanchez MI, Nardelli A, Borojevic R, De Palma G, Calo NC, McCarville J, Caminero A, Basra D, Mordhorst A, Ignatova E, Hansen S, Uhde M, Norman GL, Murray JA, Smecuol E, Armstrong D, Bai JC, Schuppan D, Collins SM, Alaedini A, Moayyedi P, Verdu EF, Bercik P. Gluten-Free Diet Reduces Symptoms, Particularly Diarrhea, in Patients With Irritable Bowel Syndrome and Antigliadin IgG. Clin Gastroenterol Hepatol. 2021 Nov;19(11):2343-2352.e8. doi: 10.1016/j.cgh.2020.08.040. Epub 2020 Aug 19. PMID 32827724